CLINICAL TRIAL: NCT06810479
Title: A Randomised, Controlled Cross Over Study Comparing Two Mandibular Advancement Devices in the Treatment of Mild-to-moderate Obstructive Sleep Apnea
Brief Title: A Study Comparing Two Mandibular Advancement Devices in the Treatment of Sleep Apnea
Acronym: MRA OSA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Z-2025010
Record Dates: First submitted 2025-01-24; First posted 2025-02-05 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-01

CONDITIONS: Apnea, Obstructive
Keywords: sleep apnea; MRA; mandibular repositioning appliance
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: randomised, controlled cross over study comparing two mandibular advancement devices
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MRA1MRA2 (Experimental): Use of MRA device 1 for 3 months, use of MRA device 2 for 3 months
  Interventions: Diagnostic Test: Polygraphy; Other: Questionaire; Other: Question
- MRA2MRA1 (Experimental): Use of MRA device 2 for 3 months, use of MRA device 1 for 3 months
  Interventions: Diagnostic Test: Polygraphy; Other: Questionaire; Other: Question

INTERVENTIONS:
Diagnostic Test: Polygraphy — Polygraphy will be caried out at the patients home to evaluate each MRA after 3 monhts
Other: Questionaire — Epworth Sleepiness Scale
  o Johns, Murray W. "A New Method for Measuring Daytime Sleepiness: The Epworth Sleepiness Scale." Sleep, vol. 14, no. 6, 1991, pp. 540-545.
Other: Questionaire — Patient experience questionnaire
  o Ng, E.T., Perez-Garcia, A., en Lagravère-Vich, M.O. "Development and Initial Validation of a Questionnaire to Measure Patient Experience with Oral Appliance Therapy." Journal of Clinical Sleep Medicine, vol. 19, nr. 8, 1 aug. 2023, pp. 1437-1445. doi: 10.5664/jcsm.10562. PMID: 37082817; PMCID: PMC10394373
Other: Question — Patient final choice of preferred MRA

SUMMARY:
The goal of this randomised, controlled cross-over study is to compare two mandibular repositioning devices (MRA) already on the market in the treatment of mild-to-moderate obstructive sleep apnea.

Patiënt will test the first MRA for 3 months, after a wash out period of 2 weeks they will test the second MRA for 3 months. It will be randomised what type of MRA will be tested first and second.

DETAILED DESCRIPTION:
A mandibular repositioning appliance (MRA) is the primary treatment option for patients with mild to moderate obstructive sleep apnea (OSA), as well as for those with severe OSA who are intolerant to continuous positive airway pressure (CPAP) therapy or for whom surgical interventions are not viable. MRAs function by advancing the mandible, thereby increasing the volume of the upper airway and reducing its tendency to collapse during sleep. Various types of MRAs are available, and multiple classification systems can be employed to distinguish between these different types.

Mandibular repositioning appliances (MRAs) can be either custom-made or universal. Custom-made devices, which are typically more expensive, are fabricated in a dental laboratory using dental impressions. In contrast, prefabricated devices, often thermoplastic MRAs, are generally less costly and readily available over the counter.

Mandibular repositioning appliances (MRAs) can be classified as non-titratable, also known as monoblock devices, which have a fixed position, or titratable devices, which allow for gradual adjustment of the mandibular position until the desired therapeutic effect is achieved. Current guidelines recommend the use of titratable MRAs.

Titratable mandibular repositioning appliances (MRAs) can be further categorized into two types: midline traction devices, where the upper and lower components are connected at the front of the device, and bilateral thrust devices, where the upper and lower components are linked in the lateral or (pre-)molar regions.

Within the latter category, various designs exist, including devices that are adjustable on both sides using Hyrax screws and 3D-printed devices equipped with a series of lower components that allow for adjustments in mandibular position.

An example of an MRA adjustable with Hyrax screws is the SomnoDent® device (SomnoMed, Denton, Texas, USA). An example of a device utilizing a series of lower components for titration is the OrthoApnea appliance (ORTHOAPNEA S.L., Málaga, Spain), which features a specific attachment mechanism.

Although studies have already been published comparing different types of "bilateral thrust" devices, no studies to date have directly compared the categories mentioned above. The hypothesis of the investigators is that both appliances have similar effectiveness in the treatment of mild-to-moderate obstructive sleep apnea.

Primary objective:

Improvement of AHI, measured by polygraphy before treatment and after treatment with each MRA.

Secondary objective;

* Peripheral oxygen saturation, measured by polygraphy before treatment and after treatment with each MRA

  * Average saturation
  * Lowest saturation
  * Oxygen desaturation index >3% (events/h)
  * Total duration with saturation < 90%
* Epworth Sleepiness Scale, taken before treatment and after treatment with each MRA
* Patient experience questionnaire, taken before treatment and after treatment with each MRA
* Patient final choice of preferred MRA

Endpoints:

The investigators assess the objective improvement in OSA by comparing polygraphy results taken before and after treatment with each MRA. To evaluate the subjective effects of the MRA, the investigators compare the scores from the Epworth Sleepiness Scale. The participants subjective experience with each MRA type is measured using a patient experience questionnaire, along with noting the final preference for device type of the participants.

Study design:

* Randomized, controlled cross-over study
* Study population: Patients referred to the Department of Oral and Maxillofacial Surgery at ZOL Genk for Mandibular Repositioning Appliance (MRA) therapy, aged 18 years or older diagnosed with an Apnea-Hypopnea Index (AHI) between 5 and 30 events per hour.

Inclusion criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Provide signed and dated informed consent
* Males or females aged 18 and above
* Apnea-Hypopnea Index (AHI) between 5 and 30 events per hour diagnosed by a polysomnography

Exclusion criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Previous surgery on the upper airways
* Prior treatment of OSA (CPAP or MRA)
* Presence of unstable cardiovascular conditions, neurological, mental, or psychiatric disorders
* Insufficient dental or periodontal condition for a mandibular repositioning appliance (MRA)
* Presence of temporomandibular joint dysfunction

ELIGIBILITY:
In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Provide signed and dated informed consent
* Males or females aged 18 and above
* Apnea-Hypopnea Index (AHI) between 5 and 30 events per hour diagnosed by a polysomnography

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Previous surgery on the upper airways
* Prior treatment of OSA (CPAP or MRA)
* Presence of unstable cardiovascular conditions, neurological, mental, or psychiatric disorders
* Insufficient dental or periodontal condition for a mandibular repositioning appliance (MRA)
* Presence of temporomandibular joint dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
AHI | 3 monthts after use of first MRA (mandibular advancement device), 3 months after use of second MRA (mandibular advancement device)
  Improvement of AHI (apnea-hypopnea index), measured by polygraphy before treatment and after treatment with each MRA. The goal of the mandibular advancement device is to reduce the number of apneas and hypopneas per hour, apneas are periods when a person stops breathing and hypopneas are instances where airflow is blocked, causing shallow breathing. This is measured by a polygraphy-test overnight at the patiënts home.

SECONDARY OUTCOMES:
Peripheral oxygen saturation 1 | 3 monthts after use of first MRA, 3 months after use of second MRA
  Measured by polygraphy
  * Average saturation (measured in %)
  * Lowest saturation (measured in %)
  Oxygen saturation in percent is the fraction of oxygen-saturated haemoglobin relative to total haemoglobin (unsaturated + saturated) in the blood * 100%
Peripheral oxygen saturation 2 | 3 monthts after use of first MRA, 3 months after use of second MRA
  Measured by polygraphy
  o Oxygen desaturation index >3% (events/h)
  Desaturation episodes are defined as a decrease in the mean oxygen saturation of ≥3% for more than 10 seconds per hour
Peripheral oxygen saturation 3 | 3 monthts after use of first MRA, 3 months after use of second MRA
  Measured by polygraphy
  o Total duration with saturation < 90%
  The percentage of cumulative time with oxygen saturation below 90% in total sleep time.
ESS | 3 monthts after use of first MRA, 3 months after use of second MRA
  Epworth Sleepiness Scale (questionaire)
  The minimum value is 0 and the maximum value is 24. A higher score means a worse outcome, indicating more excessive daytime sleepiness.
  The Epworth Sleepiness Scale is scored by adding up the individual scores for each of the eight questions. Each question is rated on a scale of 0 to 3, with 0 being "no chance of dozing" and 3 being "high chance of dozing." ter daytime sleepiness.
  Score range Interpretation 0-5 Lower normal daytime sleepiness 6-10 Normal daytime sleepiness 11-12 Mild excessive daytime sleepiness 13-15 Moderate excessive daytime sleepiness 16-24 Severe excessive daytime sleepiness
Patient experience questionnaire | 3 monthts after use of first MRA, 3 months after use of second MRA
  Patient experience questionnaire, taken before treatment and after treatment with each MRA
  Oral Appliance Therapy Patient Experience Questionnaire (OATPEQ). The minimum value is 0 and the maximum value is 100. A higher score means a better outcome, indicating a more positive patient experience with oral appliance therapy.
Final choice | after the use of each MRA for 3 months
  Patient final choice of preferred MRA.
  At the final visit, after using each MRA (type 1 and type 2) for three months (with a two-week washout period in between), the patient will choose their preferred device. The final choice will be noted down after oral questioning.

REFERENCES:
- [Background] Ng ET, Perez-Garcia A, Lagravere-Vich MO. Development and initial validation of a questionnaire to measure patient experience with oral appliance therapy. J Clin Sleep Med. 2023 Aug 1;19(8):1437-1445. doi: 10.5664/jcsm.10562. PMID 37082817
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Zhou J, Liu YH. A randomised titrated crossover study comparing two oral appliances in the treatment for mild to moderate obstructive sleep apnoea/hypopnoea syndrome. J Oral Rehabil. 2012 Dec;39(12):914-22. doi: 10.1111/joor.12006. Epub 2012 Sep 27. PMID 23016888
- [Background] Vezina JP, Blumen MB, Buchet I, Hausser-Hauw C, Chabolle F. Does propulsion mechanism influence the long-term side effects of oral appliances in the treatment of sleep-disordered breathing? Chest. 2011 Nov;140(5):1184-1191. doi: 10.1378/chest.10-3123. Epub 2011 May 26. PMID 21622552
- [Background] Shi X, Lobbezoo F, Chen H, Rosenmoller BRAM, Berkhout E, de Lange J, Aarab G. Comparisons of the effects of two types of titratable mandibular advancement devices on respiratory parameters and upper airway dimensions in patients with obstructive sleep apnea: a randomized controlled trial. Clin Oral Investig. 2023 May;27(5):2013-2025. doi: 10.1007/s00784-023-04945-z. Epub 2023 Mar 17. PMID 36928350
- [Background] Lawton HM, Battagel JM, Kotecha B. A comparison of the Twin Block and Herbst mandibular advancement splints in the treatment of patients with obstructive sleep apnoea: a prospective study. Eur J Orthod. 2005 Feb;27(1):82-90. doi: 10.1093/ejo/cjh067. PMID 15743867
- [Background] Uniken Venema JAM, Rosenmoller BRAM, de Vries N, de Lange J, Aarab G, Lobbezoo F, Hoekema A. Mandibular advancement device design: A systematic review on outcomes in obstructive sleep apnea treatment. Sleep Med Rev. 2021 Dec;60:101557. doi: 10.1016/j.smrv.2021.101557. Epub 2021 Oct 1. PMID 34662769
- [Background] Schmidt-Nowara W, Lowe A, Wiegand L, Cartwright R, Perez-Guerra F, Menn S. Oral appliances for the treatment of snoring and obstructive sleep apnea: a review. Sleep. 1995 Jul;18(6):501-10. doi: 10.1093/sleep/18.6.501. PMID 7481421
- [Background] Dieltjens M, Vanderveken O. Oral Appliances in Obstructive Sleep Apnea. Healthcare (Basel). 2019 Nov 8;7(4):141. doi: 10.3390/healthcare7040141. PMID 31717429
- [Background] Almeida FR, Lowe AA. Principles of oral appliance therapy for the management of snoring and sleep disordered breathing. Oral Maxillofac Surg Clin North Am. 2009 Nov;21(4):413-20. doi: 10.1016/j.coms.2009.07.002. PMID 19944341
- [Background] Ramar K, Dort LC, Katz SG, Lettieri CJ, Harrod CG, Thomas SM, Chervin RD. Clinical Practice Guideline for the Treatment of Obstructive Sleep Apnea and Snoring with Oral Appliance Therapy: An Update for 2015. J Clin Sleep Med. 2015 Jul 15;11(7):773-827. doi: 10.5664/jcsm.4858. PMID 26094920